CLINICAL TRIAL: NCT06047574
Title: Multidisciplinary Combined Precise Diagnosis and Treatment of Polycystic Ovary Syndrome
Brief Title: Multidisciplinary Diagnosis and Treatment of Polycystic Ovary Syndrome
Status: Recruiting | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Other Study IDs: Multidisciplinary treat PCOS
Record Dates: First submitted 2023-09-11; First posted 2023-09-21 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Clinical characteristics; New biomarkers; Multidisciplinary
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS: 1. Oligomenorrhea/amenorrhea
  2. Clinical androgen excess or biochemical androgen excess
  3. Polycystic ovary showed by gynecological ultrasound
  Interventions: Other: This study does not involve any interventions
- NOPCOS: not meet Rotterdam standards
  Interventions: Other: This study does not involve any interventions

INTERVENTIONS:
Other: This study does not involve any interventions — This study does not involve any interventions

SUMMARY:
The investigators collected clinical data and serum samples of patients with polycystic ovary syndrome (PCOS) in this study, used statistical software such as SPSS for date analysis, and used experimental techniques such as ELISA and flow cytometry to detect serum samples, aiming to explore the relationship between the body anthropometry, skin conditions, psychosomatic status, diet, sleep, exercise, glucose and lipid metabolism, gonadal hormones, and body fat distribution in patients with polycystic ovary syndrome, and to discovery new biomarkers. Multidisciplinary exploration of the mechanisms of disease occurrence and development, the establishment of a PCOS multicenter, multidisciplinary and multidimensional clinical research database, combined with the established statistical analysis strategy for big data and analysis, to promote the realization of more accurate personalized medicine.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18- 45;

Exclusion Criteria:

* Female patients younger than 18 years old or older than 45 years old;
* Ovulatory disorders caused by premature ovarian failure, pituitary amenorrhea, hypothalamic amenorrhea, and thyroid dysfunction;
* Congenital adrenal hyperplasia, reservoir Hin syndrome, hyperprolactinemia, adrenal tumors and other diseases that cause hyperandrogenism;
* Abnormal liver or renal function((≥ 3 times of the upper limit of normal range)
* Type 1 diabetes, single gene mutation diabetes, or pancreatic damage Diabetes or other secondary diabetes caused by diabetes;
* History of malignant tumors;
* Severe infection, severe anemia, neutropenia and other systemic chronic diseases;
* Undergo total hysterectomy or ovarian adnexectomy;
* Mental illness, dementia or other cognitive behavioral problems;
* Use hypoglycemic drugs that may affect insulin resistance and androgen levels in the last 3 months, including thiazolidinediones, metformin, SGLT-2, and acarbose and GLP-1RA and other drugs;
* Use letrozole, clomiphene, oral contraceptives, glucocorticoids, gonadotropins, gonadotropin-releasing hormone agonists, anti-androgens (spironolactone, Cyproterone acetate, flutamide, etc.) and other drugs for the treatment of PCOS.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Polycystic ovary syndrome (PCOS) is a common dis-order in women that is characterized by hyperandro-genism (that is, evidence of excess male hormone or androgen effect; clinically, such as hirsut-ism, and/or biochemically, such as hyperandrogen aemia or excess levels of androgen), ovulatory dysfunction (including menstrual dysfunction) and polycystic ovarian morphology (PCOM; an excessive number of preantral follicles in the ovaries).
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Fibrinogen-like-protein 1 (FGL1) | baseline
  Fibrinogen-like-protein 1 (FGL1), is a novel hepatokine that plays an important role in hepatic steatosis, insulin resistance and obesity. There is no maximum or minimum value for this parameter and the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
body mass index ,BMI | baseline
  BMI=weight(kg)/height(m)^2
Waist/hip Ratio,WHR | baseline
  WHR=Waist Circumference(cm)/Hip Circumference(cm)
Number of menstruation in the last year | baseline
  physiological parameter,the total number of menstrual periods in the last year
Ferriman-Gallwey score | Time Frame: baseline
  The minimum value of Ferriman-Gallwey score is 0 and the maximum value is 44. An Ferriman-Gallwey score greater than or equal to 6 is considered to be a clinical manifestation of androgen excess.
HOMA-IR | baseline
  Homeostatic model assessment insulin resistance index
TT | baseline
  total testosterone (nmol/L)
FT | baseline
  Free testosterone (nmol/L)
LH | baseline
  luteinizing hormone
FSH | baseline
  follicle-stimulating hormone
FBG | baseline
  fasting blood-glucose
PBG | baseline
  postprandial blood-glucose
FINS | baseline
  fasting serum insulin
PINS | baseline
  postprandial serum insulin
AST | baseline
  aspartate aminotransferase
ALT | baseline
  alanine aminotransferase
UA | baseline
  Uric acid
CR | baseline
  Creatinine
LDL-c | baseline
  low-density lipoprotein cholesterol
HDL-c | baseline
  high-density lipoprotein cholesterol
TC | baseline
  Total Cholesterol (mmol/L)
TG | baseline
  Triglyceride (mmol/L)
Interleukin 22#IL-22 | baseline
  The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Interleukin 6#IL-6 | baseline
  IL-6. The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Interleukin 8# IL-8 | baseline
  The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Tumor Necrosis Factor# TNF | baseline
  The factor reflects that the organism is in an inflammatory state. There is no maximum or minimum value for the factor and the higher scores mean a worse outcome.
Chemerin | baseline
  A adipocytokine.The factor is expressed in adipose tissue and is related to specific adipose tissue function.
omentin-1 | baseline
  A adipocytokine.The factor is expressed in adipose tissue and is related to specific adipose tissue function.
leptin | baseline
  A adipocytokine.The factor is expressed in adipose tissue and is related to specific adipose tissue function.
RBP-4 | baseline
  A adipocytokine.The factor is expressed in adipose tissue and is related to specific adipose tissue function.
adiponectin | baseline
  A adipocytokine. The factor is expressed in adipose tissue and is related to specific adipose tissue function.
DHEAS | baseline
  dehydroepiandrosterone（nmol/L）
SHBG | baseline
  sex hormone-binding globulin (nmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Shanghai 10th People's Hospital
Locations (1):
- Department of Endocrinology, Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No